CLINICAL TRIAL: NCT05184335
Title: Phase 3, Randomized, 28 Days, Double-blind, Placebo-controlled, Multicenter Study to Assess the Safety and Efficacy of Brilaroxazine (RP5063) in Subjects With Schizophrenia, Followed by a 52-Week Open-label Extension
Brief Title: Safety and Efficacy of Brilaroxazine (RP5063) in Schizophrenia
Acronym: RECOVER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Reviva Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVP-30-001 RECOVER
Record Dates: First submitted 2021-11-29; First posted 2022-01-11 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — RP5063

STUDY DESIGN:
Intervention Model Description: This is a parallel group efficacy and safety study with 3 treatment arms (2 active, one placebo, randomized 1:1:1) that is blinded for participants and involved study staff except dedicated unblinded individuals in statistics and drug safety. The OLE part will provide RP5063 15 mg, 30mg or 50mg OD open label to all participants.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RP5063 15 mg once daily (Active Comparator): administered OD for 28 days then flexibly 15-50mg over a period of 52 weeks.
  Interventions: Drug: Brilaroxazine
- RP5063 (brilaroxazine) 50 mg once daily (Active Comparator): administered OD for 28 days, then flexibly 15-50mg over a period of 52 weeks
  Interventions: Drug: Brilaroxazine
- Placebo (Placebo Comparator): administered OD for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Brilaroxazine — RP5063, a new chemical entity (NCE), is a novel multimodal neuromodulator intended for treating schizophrenia and comorbid conditions. This drug is an investigational drug and has not been approved for treatment or marketing. RP5063 belongs to a class of third generation antipsychotics called Dopamine-Serotonin System Stabilizers. The chemical name of the RP5063 active pharmaceutical ingredient (API) is 6-(4-(4-(2,3-dichlorophenyl)-piperazin-1-yl)-butoxy)-2H-benzo[b][1,4]oxazin-3(4H)-one hydrochloride.
  Other Names: RP5063
  Arms: RP5063 (brilaroxazine) 50 mg once daily; RP5063 15 mg once daily
Other: Placebo — RP5063 matching Placebo
  Arms: Placebo

SUMMARY:
This study is to evaluate the effect and safety of Brilaroxazine in patients with acute schizophrenia compared to the placebo short and long-term. Brilaroxazine will be given at fixed doses of 15 mg or 50 mg once daily over 4 weeks, then in the long-term flexible doses 15-50mg daily over a period of 52 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind (DB), placebo-controlled, multicenter study to assess the efficacy and safety of RP5063 (brilaroxazine) at fixed doses of 15 mg or 50 mg, administered once daily (OD) for 28 days (28 days DB treatment) in subjects with an acute exacerbation of schizophrenia. The study further will assess the safety of RP5063 (brilaroxazine) at flexible doses of either 15, 30 or 50 mg administered OD in an Open Label (OL) treatment over a period of 52 weeks (52-week OL treatment part), in subjects with stable schizophrenia. The OL treatment will have 2 populations of stable schizophrenia: DB rollover and de novo subjects.

The study comprises 2 parts: a 28-day DB treatment, followed by 52 weeks OL treatment.

The total duration of the study is 56 weeks (28 days/4 weeks DB treatment and 52-weeks OL treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, aged 18 to 65 years
2. Subject reads, understands, and signs an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved current ICF prior to performing any of the Screening procedures
3. Diagnosis schizophrenia

Exclusion Criteria:

1. Has a history of treatment resistance exhibited by any of the following:

   1. No or minimal response to at least 2 periods of treatment lasting 28 days or longer, with antipsychotic agents at the maximally tolerated dose.
   2. Lifetime history of clozapine use
   3. History of electroconvulsive therapy (ECT) for treatment of schizophrenia within the past 5 years.
2. Is treatment-naïve for schizophrenia.
3. Primary current diagnosis other than schizophrenia or a comorbid diagnosis that is primarily responsible for the current symptoms and functional impairment.
4. Has a current diagnosis of a psychotic disorder other than schizophrenia or a behavioral disturbance thought to be due to substance abuse disorder.
5. Meets criteria for moderate-to-severe substance use disorder within past 6 months prior to Screening (excluding those related to caffeine or nicotine).
6. Has a history of the following: (a) traumatic brain injury causing ongoing cognitive difficulties, Alzheimer's disease, or another form of dementia, or any chronic organic disease of the central nervous system (CNS) (b) intellectual disability of a severity that would impact ability to participate in the study.
7. Subject has a current primary DSM-5 diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, post-traumatic stress disorder, obsessive-compulsive disorder, manic episode, hypomania, panic disorder, delirium, amnestic or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
8. On antipsychotic within the Screening Period (minimum 3 days prior to Baseline and throughout the study).
9. Within 28 days prior to Baseline: monoamine oxidase (MAO) inhibitors, CNS stimulants, potent CYP3A4/5 enzyme-inducing drugs including but not limited to rifampin and carbamazepine and strong CYP3A4/5 inhibitors like ketoconazole, itraconazole, clarithromycin, etc. (see Appendix 20.1 for prohibited medications).
10. Antipsychotic depot medication within 5 half-lives prior to Baseline.
11. Positive Urine Drug Screen for drugs of abuse, including amphetamines, barbiturates, cocaine, ecstasy, phencyclidine or opiates meeting criteria of moderate-to-severe DSM-5 substance use disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Double Blind Safety and Efficacy of Brilaroxazine (RP5063) | 28 days
  decrease in Positive and Negative Symptoms Assessment total score compared to placebo from Baseline to Day 28.
Open label Safety and Efficacy of Brilaroxazine (RP5063) | 52 weeks
  (brilaroxazine) tablets (at flexible doses of 15 mg or 30 mg 0r 50mg OD) in an treatment part over a period of 52 weeks in stable schizophrenia subjects. The endpoints would be incidence of Treatment-Emergent Adverse Events [Safety and Tolerability])

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Reviva Pharma
Locations (17):
- United States (17):
  - Reviva site, Phoenix, Arizona
  - Reviva site, Bentonville, Arkansas
  - Reviva site, Little Rock, Arkansas
  - Reviva site, Rogers, Arkansas
  - Reviva site, Garden Grove, California
  - Reviva site, Lemon Grove, California
  - Reviva site, Riverside, California
  - Reviva site, Hollywood, Florida
  - Reviva site, Miami Lakes, Florida
  - Reviva site, Atlanta, Georgia
  - Reviva site, Decatur, Georgia
  - Reviva site, Chicago, Illinois
  - Reviva site, Gaithersburg, Maryland
  - Reviva site, Boston, Massachusetts
  - Reviva site, Oklahoma City, Oklahoma
  - Reviva site, Austin, Texas
  - Reviva site, Richardson, Texas